CLINICAL TRIAL: NCT03471221
Title: Psychological Benefits and Potential Pathogen Transmission in Hospitalized Pediatric Oncology Patients Receiving Therapy Dog Visits: a Randomized Controlled Trial
Brief Title: Helping Improve Pediatric Patient Outcomes
Acronym: HIPPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1R21HD091877 (NIH)
Record Dates: First submitted 2018-02-16; First posted 2018-03-20 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pediatric Cancer, Animal-Assisted Activities
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes Assessors include clinical research assistants and laboratory personnel. Laboratory personnel will be blinded. Clinical research assistants collecting surveys and specimens will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy Dog Visits (Experimental): Participants randomized to Therapy Dog Visits will receive a visit from a therapy dog and handler team up to one time per week for up to four weeks, depending on length of hospitalization and therapy dog team capacity.
  Therapy dog visits will last up to about 20 minutes and activities may include: petting the dog, watching the dog perform a trick, and talking with the dog handler.
  All activities will follow the current procedures and regulations in place at Seattle Children's Hospital.
  Interventions: Behavioral: Therapy Dog Visit
- Control Group (No Intervention): Participants randomized to the Control Group will receive usual medical care.

INTERVENTIONS:
Behavioral: Therapy Dog Visit — Animal Assisted Activities (AAA) provide opportunities for motivational, educational, recreational, and/or therapeutic benefits to enhance quality of life. AAA are delivered in a variety of environments by specially trained professionals, paraprofessionals, and/or volunteers, in association with animals that meet specific criteria.
  Key features of AAA are as follows:
  1. Specific treatment goals are not planned for each visit.
  2. Volunteers and treatment providers are not required to take detailed notes.
  3. Visit content and activities are spontaneous.
  4. Visit length can be as long or as short as needed.
  Other Names: Animal-Assisted Activities
  Arms: Therapy Dog Visits

SUMMARY:
This study involves two distinct activities:

The first is a randomized controlled trial (RCT) to assess the efficacy and safety of therapy dog visits for children with cancer. This activity has the following specific objectives:

1. To assess the effect of therapy dog visits on psychosocial outcomes and satisfaction with care among pediatric oncology inpatients.
2. To determine whether therapy dog visits increase microbial levels on children's hands.

The Investigators hypothesize that therapy dog visits will reduce patient distress, lower treatment-related anxiety, increase happiness, and improve satisfaction with hospital care. The Investigators further hypothesize that therapy dog visits (including standard hand sanitization) will not increase microbial levels on children's hands.

Once the main study aims for the first study activity have been completed, the research study team will begin recruitment for the second activity. The second activity is an observational study to describe microbial levels before a dog visit, after a dog visit but before hand cleaning, and after hand cleaning. This phase will provide additional information for Aim 2 that cannot be obtained during the RCT given the nature of the RCT design. The Investigators will proceed with the observational study only if all main study activities can be completed within the study timeline.

DETAILED DESCRIPTION:
This study tests whether therapy dog visits reduce distress, lower treatment-related anxiety, increase happiness, and improve satisfaction with hospital care, and whether these visits transmit pathogens.

The first activity is a randomized controlled trial (RCT) in which patients will be randomized to either the intervention (therapy dog visits) or control (usual care). All patients will complete a baseline survey and hand sampling (i.e., removal of materials of hands via use of liquid inside a glove) and answer questions from study staff (e.g., about pets at home, which hand is dominant) before randomization. Parents will also complete a baseline survey. Patients in the intervention group will receive therapy dog visits. At the first therapy dog visit after enrollment, the research study team will collect visit-level psychosocial measures and perform hand sampling. Similar procedures will be performed on usual care patients. Patients in the intervention group will receive subsequent dog visits ~1x/week for up to 4 weeks if there sufficient dog team capacity. At hospital discharge, ~3 days post-discharge and 9 weeks post-discharge, the research study team will administer surveys to patients and their parents in both groups.

Informed consent/assent will be performed for patients who agree to participate in the study and preliminarily meet eligibility criteria. The parent/legal guardians of participants who are enrolled in will be approached for their informed consent to complete surveys. After informed consent/assent has been obtained, baseline surveys will be administered and hand samples will be collected. The study staff will then assess the patient's ability to tolerate and willingness to perform future psychological assessments and hand samplings. Patients willing to proceed with the study will be randomized to either the intervention arm (visits from a therapy dog) or the control arm (no visits from a therapy dog). Participants will be randomized (1:1) to each group and stratified by age (≥13 vs <13 years). Participants will maintain their randomization assignment during any subsequent hospitalizations that occur during their participation in the study.

The second activity is an observational study of patients receiving therapy dog visits that will provide additional information on microbial levels. The observational study which involves a one-time therapy dog visit. Children will be instructed to touch the dog with both hands. Both hands will be sampled before the visit. A randomly selected hand will be sampled immediately after the visit (before hand sanitization). The other hand will be sampled after sanitization.

ELIGIBILITY:
Inclusion Criteria:

English-speaking patients aged 5-17 years who have been admitted to the Seattle Children's Hospital Cancer Care Unit and who are on the oncology service irrespective of specific oncologic diagnosis, sex, race, and ethnicity.

Exclusion Criteria:

Are allergic to dogs or have a sensitivity to dogs; Are afraid of dogs; Are on the bone marrow transplant service; Have isolation precautions in place per Infection Prevention policies (e.g. viral respiratory precautions, contact precautions, etc.); Skin on hands not intact (e.g. moderate to severe eczema involving the hands or other generalized skin breakdown); Have no English-speaking parent/legal guardian; Have no parent/legal guardian able to provide written consent; For observational study, unwilling or unable to pet the dog with both hands.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) total distress score | Immediately after first visit (Intention to Treat)
  The PedsQL VAS total score is a measure of present or in-the-moment distress. It is computed as the average of 6 scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt). Each scale ranges from 0-100, with lower scores indicating lower distress. For the overall score, lower values indicate lower total distress.
Microbial load (colony forming units; cfu) on child hands | Immediately after first visit (Intention to Treat and Per Protocol)
  Microbial load on child hands

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) total distress score | Immediately after first visit (Per Protocol)
  The PedsQL VAS total score is a measure of present or in-the-moment distress. It is computed as the average of 6 scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt). Each scale ranges from 0-100, with lower scores indicating lower distress. For the overall score, lower values indicate lower total distress.
Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) individual scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt) | Immediately after first visit (Intention to Treat)
  Each of 6 scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt) ranges from 0-100, with lower scores indicating a better outcome.
Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) emotional distress summary score. | Immediately after first visit (Intention to Treat)
  The PedsQL VAS emotional distress summary score is a measure of present or in-the-moment emotional distress. It is computed as the average of 4 scales (afraid/scared, sad/blue, angry, worry). Each scale ranges from 0-100, with lower scores indicating lower distress. For the overall score, lower values indicate lower emotional distress.
Presence of Clinically Important Organisms | Immediately after first visit (Intention to Treat and Per Protocol)
  The presence of each of the following nine organisms:
  Staphylococcus aureus (further evaluated for methicillin-resistance); Vancomycin-resistant enterococci; Malassezia; Aspergillus; Pasteurella; Enterobacteriaceae (further assessed for multidrug resistance); Acinetobacter (further assessed for multidrug resistance); Pseudomonas aeruginosa (further assessed for multidrug resistance); Clostridium difficile
Pediatric Quality of Life Inventory (PedsQL) Cancer Module: treatment anxiety dimension | Hospital discharge (hospital discharge date varies by patient), 3 days post-hospital discharge, and 9-weeks post-hospital discharge, (Intention to Treat)
  Treatment anxiety is one dimension measured within the PedsQL Cancer Module. It consists of 3 questions on a Likert scale. Items are reversed scored and linearly transformed on a 0-100 scale and then averaged. Higher scores indicate lower treatment anxiety.
Patient feelings when thinking about being in the hospital (afraid/scared, sad/blue, angry; worried) | Hospital discharge (hospital discharge date varies by patient), 3 days post-hospital discharge, and 9-weeks post-hospital discharge), (Intention to Treat)
  Each feeling (afraid/scared, sad/blue, angry, worried) is measured as either, not present, a little bit present, present, or strongly present.
The Positive and Negative Affect Schedule (PANAS): parent measure of child's positive affect | Primary: Hospital discharge (hospital discharge date varies by patient); secondary: 3 days post-hospital discharge and 9-weeks post-hospital discharge (Intention to Treat)
  The parent report of the child's positive affect consists of 5 positive feelings/emotions each scored on a 5-point Likert scale. Low scores represent worse outcomes. The total score (range: 5-25) is obtained by summing the items.
The Positive and Negative Affect Schedule (PANAS): parent measure of child's negative affect | Primary: Hospital discharge (hospital discharge date varies by patient); secondary: 3 days post-hospital discharge and 9-weeks post-hospital discharge (Intention to Treat)
  The parent report of the child's negative affect consists of 5 negative feelings/emotions each scored on a 5-point Likert scale. Low scores represent better outcomes. The total score (range: 5-25) is obtained by summing the items.
Six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI) | Immediately after first visit, (Intention to Treat)
  The short form of the Spielberger State-Trait Anxiety scale will be used to measure parent anxiety. It consists of six items, each on a 4-point Likert scale. The total score is obtained by reverse scoring the three positive items, summing the six scores together, and then multiplying by 20/6. Total scores range from 20 to 80 with higher numbers representing worse outcomes.
Parent rating of hospital | Primary: Hospital discharge (hospital discharge date varies by patient); secondary: 3 days post-hospital discharge and 9-weeks post-hospital discharge (Intention to Treat)
  Parents rate the hospital on a 11-point Likert scale. Scores range from 0 to 10. Lower scores represent worse hospital ratings.
Microbial load (colony forming units; cfu) on hands that touched the dog versus hands of medically eligible controls | Immediately after first visit
  Microbial load on hands that touched the dog versus hands of medically eligible controls

OTHER OUTCOMES:
Change in microbial load (colony forming units; cfu) on hands that touched the dog | Immediately before and immediately after first visit
  Microbial load change from pre-visit to post-visit in the intervention group; only among participants who got a dog visit and only the hand(s) that touched the dog.
Infections | From enrollment through 1-month post-completion of participation (participation = up to 4-weeks post-enrollment).
  Counts of persons and Infections/Positive Cultures, including descriptions
Change in Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) total score among patients receiving a therapy dog visit | Immediately before and immediately after first visit
  Score change from pre-visit to post-visit. The PedsQL VAS total score is a measure of present or in-the-moment distress. It is computed as the average of 6 scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt). Each scale ranges from 0-100, with lower scores indicating lower distress. For the overall score, lower values indicate lower total distress. Score changes can range from -100 to 100. Negative changes in scores indicate better outcomes. Intervention Group only and only participants who received a dog visit.
Change in Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) emotional distress summary score among patients receiving a therapy dog visit | Immediately before and immediately after first visit
  Score change from pre-visit to post-visit. The PedsQL VAS emotional distress summary score is a measure of present or in-the-moment emotional distress. It is computed as the average of 4 scales (afraid/scared, sad/blue, angry, worry). Each scale ranges from 0-100, with lower scores indicating lower distress. For the overall score, lower values indicate lower emotional distress. Score changes can range from -100 to 100. Negative changes in scores indicate better outcomes. Intervention Group only and only participants who received a dog visit.
Change in Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) individual scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt) among patients receiving a therapy dog visit | Immediately before and immediately after first visit
  Individual item change from pre-visit to post-visit. Each of 6 scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt) ranges from 0-100, with lower scores indicating a better outcome. Score changes can range from -100 to 100. Negative changes in scores indicate better outcomes. Intervention Group only and only participants who received a dog visit.
Pediatric Quality of Life Inventory Present Functioning Visual Analogue Scales (PedsQL VAS) total score stratified by age | Immediately after first visit, (Intention to Treat), Stratified by Age
  The PedsQL VAS total score is a measure of present or in-the-moment distress. It is computed as the average of 6 scales (afraid/scared, sad/blue, angry, worry, tired, pain/hurt). Each scale ranges from 0-100, with lower scores indicating lower distress. For the overall score, lower values indicate lower total distress.
Pediatric Quality of Life Inventory (PedsQL) Cancer Module | Hospital discharge (hospital discharge date varies by patient, 3 days post-hospital discharge, and 9-weeks post-hospital discharge), (Intention to Treat)
  The PedsQL Cancer Module measures quality of life in children and teens with cancer based on 8 dimensions (pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance, and communication). Items are reversed scored and linearly transformed on a 0-100 scale and then summed and divided by the number of items answered. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Chubak J, Adler A, Bobb JF, Hawkes RJ, Ziebell RA, Pocobelli G, Ludman EJ, Zerr DM. A Randomized Controlled Trial of Animal-assisted Activities for Pediatric Oncology Patients: Psychosocial and Microbial Outcomes. J Pediatr Health Care. 2024 May-Jun;38(3):354-364. doi: 10.1016/j.pedhc.2023.09.010. Epub 2023 Nov 4. PMID 37930283